CLINICAL TRIAL: NCT03775122
Title: Transcutaneous Acupoint Electrical Stimulation Improve the Function of Respiration and Circulation on Elderly Patients Undergoing Colonoscopy Procedure：A Randomized-controlled Trial
Brief Title: TAES Improve the Function of Respiration and Circulation on Elderly Patients Undergoing Colonoscopy Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: renji-2018-074
Record Dates: First submitted 2018-12-10; First posted 2018-12-13 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Respiratory Depression
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 sedation group (Placebo Comparator): Elderly patients under colonoscopy with sedation, but no real TAES neiguan(pc6)
  sedation is using the typical protocol for the following: Slowly peripheral intravenous injection(0.5ml/s) of fentanyl 50μg, then followed with 1.5-2.5mg/kg propofol until loss of eyelash reflex, the Observer's Assessment of Alertness/Sedation Scale (OAAS) score Level3-5.
  Interventions: Device: TAES
- Group 2 sedation+TAES group (Experimental): Elderly patients under colonoscopy both have TAES neiguan(pc6) and sedation.
  sedation is begun followed TAES. sedation is same as group2 do. TAES is same as group3 do.
  Interventions: Device: TAES

INTERVENTIONS:
Device: TAES — TAES over acupuncture point neiguan (pericardium 6) for 20min, placebo group only stick the stimulate electrode but no frequency and intensity

SUMMARY:
To explore the effectiveness of transcutaneous acupuncture electrical stimulation (TAES), a non-invasive modality in improvement of the function of respiration and circulation on elder patient during colonoscopy.

DETAILED DESCRIPTION:
To assess the function of respiratory and circulation before precondition, during colonoscopy and end of the procedure, blood cortisol and catecholamine levels were measured also.The incidence of airway support, application of vasoactive drug or atropine during procedure were recorded in the meantime.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 65 or older
2. American Society of Anesthesiologists (ASA) grade I~II
3. consent and voluntary participation in this experiment
4. patients under colonoscopy
5. none allergic to propofol and fentanyl
6. airway assessment for none difficult airway

Exclusion Criteria:

1. Allergic to propofol, fentanyl.
2. ASA is greater than or equal to grade 3
3. Abnormal respiratory tract may cause severe respiratory obstruction
4. unsatisfactory control of hypertension, systolic pressure over 160 millimeter of mercury (mmHg) or diastolic pressure over 100 mmHg
5. Hypotension, systolic pressure below 90 mmHg, heart rate (HR) <50bpm or >100bpm

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-15 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of oxygen saturation | from 20min before lay down to 24hours after performance
  The percentage of oxygen saturation between the sedation alone and sedation+TAES have at least 2 difference

CONTACTS AND LOCATIONS:
Overall Officials: Yu Weifeng, Dr, Study Director — Renji Hospital,School of Medicine,Shanghai Jiaotong University
Locations (1):
- Diansan Su, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Y, Gong Y, Huai X, Gu X, Su D, Yu W, Xie H. Effects of transcutaneous electrical acupuncture point stimulation on peripheral capillary oxygen saturation in elderly patients undergoing colonoscopy with sedation: a prospective randomized controlled trial. Acupunct Med. 2021 Aug;39(4):292-298. doi: 10.1177/0964528420960479. Epub 2020 Nov 30. PMID 33256456